CLINICAL TRIAL: NCT05697471
Title: Far Eastern Memorial Hospital
Brief Title: Comparisons of the Therapeutic Effects of Dienogest and Danazol on Endometriosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111207-F
Record Dates: First submitted 2023-01-01; First posted 2023-01-26 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — dienogest; Danazol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dienogest (Experimental)
  Interventions: Drug: Dienogest
- Danazol (Active Comparator)
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Dienogest — Dienogest 2 mg per day
  Arms: Dienogest
Drug: Danazol — Danzol 200MG per day
  Arms: Danazol

SUMMARY:
The aim of this study is to evaluate the efficacy between dienogest and danazol.

DETAILED DESCRIPTION:
Objective: Women with adenomyosis or endometripsis are often suffered from dysmenorrhea or menorrhagia. Dienogest and danazol are frequently used for the treatment of endometriosis. However, there was no literature mentioned about which medication is better for the treatment of endometriosis. Thus, the aim of this study is to evaluate the efficacy between dienogest and danazol.

Methods: All consecutive women, who have endometriosis, will be randomized to receive dienogest or danazol treatment, and will assess symptoms severity, receive CA125 examination, sonographic examination at baseline, 4 weeks and 16 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* > 20 years old
* Have an endometriosis-related condition (including adenomyosis, adenomyoma, ovarian endometrioma, or pelvic endometriosis).

Exclusion Criteria:

* Minors.
* Have a history of breast cancer or other cancers.
* Patients with vascular obstruction such as stroke.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of severity in dysmenorrhea | 16 weeks
  Between-group difference in the score of global response assessment of dysmenorrhea

SECONDARY OUTCOMES:
The change of severity in urinary symptoms | 16 weeks
  Between-group difference in the score of UDI-6
The change of severity in quality of life related to urinary symptoms | 16 weeks
  Between-group difference in the score of IIQ-7
The change of severity in menstrual amount | 16 weeks
  Between-group difference in the score of global response assessment of menstrual amount

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No